CLINICAL TRIAL: NCT00212940
Title: Increasing Patient Adherence to HIV Medications: A Prospective Intervention Study
Brief Title: Supportive Therapy for Adherence to ART(STAART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Ontario HIV Treatment Network (Network)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1999565-01H; CIHR app# 1262000 ICE:
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-07-26 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: Treatment Naive; HIV
MeSH Terms: conditions — HIV Infections | interventions — Palliative Care

INTERVENTIONS:
Behavioral: Supportive Therapy for Adherence to ART (behavior)

SUMMARY:
The purpose of this study is to determine whether a psycho-educational intervention can help people living with HIV handle the changes of treatment adherence.

DETAILED DESCRIPTION:
Participants will be randomly assigned to one of two study groups:

* Group 1: participants in this group will engage in weekly psycho-educational sessions with an HIV therapist for four weeks prior to starting their regimens. The sessions will cover topics such as becoming active in treatment care, improving coping abilities and developing skills for treatment adherence. They will also involve questionnaires and readings.
* Group 2 (the control group):participants in this group will simply receive their regular treatment regimens.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* have viral load above 500 copies/ml
* not be currently on HAART
* be able to read and speak English/French

Exclusion Criteria:

* current Substance Abuse
* actively psychotic or suicidal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2000-10; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
psycho-educational intervention can help people living with HIV handle the changes of treatment adherence

CONTACTS AND LOCATIONS:
Overall Officials: William Cameron, MD, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital, General Campus, Ottawa, Ontario, Canada